CLINICAL TRIAL: NCT01657123
Title: Effect of Hydrocortisone Stress Dose on Exercise Capacity and Post-exercise Recovery in Patients With Addison's Disease
Brief Title: Exercise Capacity and Recovery in Addison's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Smans, drs, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33088
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Addison's Disease
Keywords: exercise capacity; Addison's disease
MeSH Terms: conditions — Addison Disease | interventions — Ergometry

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Other: ergometry
- hydrocortisone stress dosage (Experimental)
  Interventions: Other: ergometry

INTERVENTIONS:
Other: ergometry — ergometry measurements
  Arms: placebo
Other: ergometry — Ergometry measurements
  Arms: hydrocortisone stress dosage

SUMMARY:
Exposure to stress alters the activity of the adrenomedullary, adrenocortical and sympathetic nervous system, depending on the type and intensity of the stressor. Physical exercise represents a stress condition influencing many systems in the body. Given a workload of at least 70-85% of Vo2max, exercise is a potent stimulus of the hypothalamic-pituitary-adrenal (HPA)-axis. The increased endogenous cortisol secretion results in important metabolic and cardiovascular effects to maintain cellular and organ homeostasis. Patients with Addison's disease are not able to meet the increased demand of adrenal steroids in case of physical exercise, which may result in an impaired exercise capacity and a prolonged post-exercise recovery. We hypothesize that a hydrocortisone stress dose increases exercise capacity and improves post-exercise recovery in patients with Addison's disease.

ELIGIBILITY:
Inclusion Criteria:

* Addison's disease
* 18-50 years
* stable glucocortiocid replacement therapy

Exclusion Criteria:

* Presence of intercurrent (acute) infectious disease
* Mental impairment (major depressive, anxiety, panic, adjustment, bipolar, psychotic, posttraumatic or borderline personality disorder)
* Presence of the following chronic diseases: diabetes mellitus, chronic obstructive pulmonary disease, renal failure, chronic anaemia, malignancy, rheumatoid arthritis
* Presence of the following cardiovascular conditions: unstable angina pectoris, history of myocardial infarction, uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise, symptomatic (severe) aortic stenosis, uncontrolled symptomatic heart failure, acute myocarditis or pericarditis, left main coronary stenosis, moderate stenotic valvular heart disease, tachyarrhythmias or bradyarrhythmias, hypertrophic cardiomyopathy and other forms of outflow tract obstruction, high-degree atrioventricular block
* History of pulmonary embolus or pulmonary infarction
* Known aortic aneurysm
* Severe hypertension (>170/100 mm Hg)
* Medication that affects cardiovascular function (beta-blocker, calcium antagonist, ACE-inhibitors, aldosterone-antagonists)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
exercise capacity | 140 minutes
  power in Watt and duration in minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands